

## STATISTICAL ANALYSIS PLAN

A Phase 1/2 open-label, multi-center, safety, preliminary efficacy and pharmacokinetic (PK) study of isatuximab (SAR650984) in combination with atezolizumab or isatuximab alone in patients with advanced malignancies

#### SAR650984-ACT15377

| STATISTICIAN: | | |
|-----------------------------|------------------------|----|
| Statistical Project Leader: | | |
| DATE OF ISSUE: 12-Sep-2019 | | |
| | Total number of pages: | 48 |

Any and all information presented in this document shall be treated as confidential and shall remain the exclusive property of Sanofi (or any of its affiliated companies). The use of such confidential information must be restricted to the recipient for the agreed purpose and must not be disclosed, published or otherwise communicated to any unauthorized persons, for any reason, in any form whatsoever without the prior written consent of Sanofi (or the concerned affiliated company); 'affiliated company' means any corporation, partnership or other entity which at the date of communication or afterwards (i) controls directly or indirectly Sanofi, (ii) is directly or indirectly controlled by Sanofi, with 'control' meaning direct or indirect ownership of more than 50% of the capital stock or the voting rights in such corporation, partnership or other entity

According to template: QSD-002643 VERSION 7.0 (20-FEB-2019)

## **TABLE OF CONTENTS**

| STATIS | TICAL ANALYSIS PLAN | 1 |
|---|---|---|
| TABLE | OF CONTENTS | 2 |
| LIST OI | ABBREVIATIONS AND DEFINITION OF TERMS | 5 |
| 1 | OVERVIEW AND INVESTIGATIONAL PLAN | |
| 1.1 | STUDY DESIGN AND RANDOMIZATION | |
| 1.1.1<br>1.1.1.1<br>1.1.1.2 | Phase 1 (safety run-in) | 7 |
| 1.1.1.3 | Maximum tolerated dose and recommended Phase 2 dose | |
| 1.1.2 | Phase 2 (efficacy signal search with a 2-stage design in each cohort) | 8 |
| 1.2 | OBJECTIVES | 9 |
| 1.2.1 | Primary objectives | 9 |
| 1.2.2 | Secondary objectives | 10 |
| 1.3 | DETERMINATION OF SAMPLE SIZE | 10 |
| 1.4 | STUDY PLAN | 11 |
| 1.5 | MODIFICATIONS TO THE STATISTICAL SECTION OF THE PROTOCOL | 11 |
| 1.6 | STATISTICAL MODIFICATIONS MADE IN THE STATISTICAL ANALYSIS PLAN | 11 |
| 2 | STATISTICAL AND ANALYTICAL PROCEDURES | 12 |
| 2.1 | ANALYSIS ENDPOINTS | 12 |
| 2.1.1 | Demographic and baseline characteristics | 12 |
| 2.1.2 | Prior or concomitant medications (other than anticancer therapies) | 14 |
| 2.1.3<br>2.1.3.1<br>2.1.3.2<br>2.1.3.3 | Efficacy endpoints Primary efficacy endpoint(s) Secondary efficacy endpoint(s) Exploratory efficacy endpoint(s) | 14<br>15 |
| 2.1.4<br>2.1.4.1 | Safety endpoints Dose limiting toxicities (DLTs) | |
| 2.1.4.1 | Adverse events variables | |
| 2.1.4.3 | Infusion associated reactions | |
| 2.1.4.4<br>2.1.4.5 | Deaths | |
| 2.1.4.5 | Vital signs variables | |

| 2.1.4.7<br>2.1.4.8<br>2.1.4.9 | Electrocardiogram variables Clinical safety laboratory assessments Immunogenicity variables | 20 |
|---|---|---|
| 2.1.5 | Pharmacokinetic variables | |
| 2.1.6.1<br>2.1.6.2<br>2.1.6.3<br>2.1.6.4 | Biomarker endpoints Microsatellite instability PD-L1 expression singleplex IHC Cluster of differentiation 38 (CD38) expression singleplex IHC Immune cell subpopulation tumor infiltration and markers co-expression multiplex immunofluorescence | 23<br>23<br>23 |
| 2.1.7 | Further therapy after discontinuation of investigational medicinal product administration during the study | |
| 2.2 | DISPOSITION OF PATIENTS | 24 |
| 2.2.1 | Randomization and drug dispensing irregularities | 25 |
| 2.3 | ANALYSIS POPULATIONS | 25 |
| 2.3.1 | All-treated population | 25 |
| 2.3.2 | DLT-evaluable population | |
| 2.3.3 | Pharmacokinetic population | |
| 2.3.4 | Biomarker Population | |
| 2.3.5 | Immunogenicity population | |
| 2.3.6 | Response evaluable population | |
| 2.4 | STATISTICAL METHODS | 26 |
| 2.4.1 | Demographics and baseline characteristics | 26 |
| 2.4.2 | Prior or concomitant medications (other than anticancer therapies) | |
| 2.4.3 | Anticancer therapies | |
| 2.4.4 | Extent of investigational medicinal product exposure and compliance | |
| 2.4.4.1 | Extent of investigational medicinal product exposure | |
| 2.4.4.2 | Isatuximab exposure | 28 |
| 2.4.4.3 | Atezolizumab exposure | 29 |
| 2.4.5 | Analyses of efficacy endpoints | |
| 2.4.5.1 | Analysis of primary efficacy endpoint(s) | |
| 2.4.5.2 | Analyses of secondary efficacy endpoints | |
| 2.4.5.3<br>2.4.5.4 | Analyses of exploratory efficacy endpoints | |
| 2.4.6 | Analyses of SI To (Phase 1 anh) | |
| 2.4.6.1<br>2.4.6.2 | Analyses of DLTs (Phase 1 only) | |
| 2.4.6.3 | Deaths | |
| 2.4.6.4 | Analyses of laboratory variables | |
| 2.4.6.5 | Analyses of vital sign variables | |
| 2.4.6.6 | Analyses of electrocardiogram variables | |

| 2.4.6.7 | Analysis of Immunogenicity | 36 |
|---|---|---|
| 2.4.7 | Analyses of pharmacokinetic variables | 36 |
| 2.4.7.1 | Cycle 1 non-compartmental analysis of isatuximab: following the 1st administration | |
| 2.4.7.2 | Over treatment concentrations: Ctrough and Ceoi of isatuximab and atezolizumab | |
| 2.4.7.3<br>2.4.7.4 | Immunogenicity impact on PK Over treatment: population PK approach of isatuximab and atezolizumab | |
| 2.4.8 | Analyses of biomarker variables | |
| 2.4.9 | Analyses of quality of life/health economics variables | 38 |
| 2.4.10 | Further therapy after discontinuation of investigational medicinal product administration during the study | 38 |
| 2.5 | DATA HANDLING CONVENTIONS | 38 |
| 2.5.1 | General conventions | 38 |
| 2.5.2 | Data handling conventions for secondary efficacy variables | 38 |
| 2.5.3 | Missing data | 38 |
| 2.5.4 | Windows for time points | 42 |
| 2.5.5 | Unscheduled visits | 42 |
| 2.5.6 | Pooling of centers for statistical analyses | 42 |
| 2.5.7 | Statistical technical issues | 42 |
| 3 | INTERIM ANALYSIS | 43 |
| 4 | DATABASE LOCK | 44 |
| 5 | SOFTWARE DOCUMENTATION | 45 |
| 6 | REFERENCES | 46 |
| 7 | LIST OF APPENDICES | 47 |
| APPENI | DIX A GENERIC RANGES FOR HEMATOLOGICAL AND BIOCHEMISTRY PARAMETERS | 48 |

## LIST OF ABBREVIATIONS AND DEFINITION OF TERMS

ADA: anti-drug antibodies ADI: actual dose intensity

AEs: adverse events

AESI: adverse events of special interest

AFP: alpha-fetoprotein

ALT: alanine aminotransferase AST: aspartate aminotransferase ATC: anatomic therapeutic category

AUC: area under the curve BOR: best overall response BUN: blood urea nitrogen

CD38: cluster of differentiation 38

CR: complete response
DCR: disease control rate
DLT: dose limiting toxicity
DoR: duration of response
ECG: electrocardiogram

ECOG: eastern cooperative oncology group

eCRF: electronic case report form EOC: epithelial ovarian cancer

EOT: end of treatment

GBM: glioblastoma multiforme
GCIG: gynaecologic cancer intergroup
HCC: hepatocellular carcinoma
IAR: infusion associated reaction
IMP: investigational medicinal product
INR: international normalized ratio

iRANO: immunotherapy response assessment in neuro-oncology

iRECIST: modified response evaluation criteria in solid tumors for immune-based

therapies

IV: intravenous

LDH: lactate dehydrogenase

MDRD: modified diet in renal disease

MedDRA: medical dictionary for regulatory activities

MTD: maximum tolerated dose

NIMP: non-investigational medicinal product

OS: overall survival

PCSA: potentially clinically significant abnormality

PFS: progression-free survival

PFS-6: progression free survival rate at 6 months

PK: pharmacokinetic PR: partial response PT: preferred term

PTT: partial thromboplastin time

Q3W: once every 3 weeks

QW: once weekly

RANO: response assessment in neuro-oncology

RBC: red blood cell

RDI: relative dose intensity

RECIST: response evaluation criteria in solid tumors

ROI: region of interest

RP2D: recommended phase 2 dose

RR: response rate

SAEs: serious adverse events

SCCHN: squamous cell carcinoma of the head and neck

SD: stable disease SOC: system organ class

TEAE: treatment-emergent adverse event TSH: thyroid stimulating hormone

TTP: time to progression TTR: time to response

WHO-DD: world health organization-drug dictionary

## 1 OVERVIEW AND INVESTIGATIONAL PLAN

## 1.1 STUDY DESIGN AND RANDOMIZATION

This is a Phase 1/2 open-label, non-randomized, multi-center, safety, preliminary efficacy, and PK study of isatuximab in combination with atezolizumab, or isatuximab alone in participants with advanced malignancies. The study will be conducted in 2 phases.

## 1.1.1 Phase 1 (safety run-in)

Participants with hepatocellular carcinoma (HCC), squamous cell carcinoma of the head and neck (SCCHN), epithelial ovarian cancer (EOC), or glioblastoma multiforme (GBM) will be enrolled in Phase 1.

## 1.1.1.1 Starting dose and de-escalation design

Starting dose is isatuximab given 10 mg/kg once weekly (QW) for 3 weeks followed by once every 3 weeks (Q3W) with atezolizumab at 1200 mg once every 3 weeks (Q3W). Dose de-escalation will be performed if necessary as defined in Table 1 below:

 Dose level (DL)
 Isatuximab
 Atezolizumab

 Starting dose
 10 mg/kg
 1200 mg

 QW × 3 ->Q3W
 Q3W

 Minus -1
 5 mg/kg
 1200 mg

 (DL-1)
 QW × 3 ->Q3W
 Q3W

Table 1 - Dose modification for Phase 1

Abbreviations: DL: Dose level; QW: once weekly, Q3W: once every 3 weeks.

At the starting dose, up to approximately 8 patients will be treated and decision will be based on the DLTs assessed in the first 6 DLT-evaluable participants (1 cycle, 21 days):

- If ≤1/6 participant has DLT, the starting dose will be the recommended Phase 2 dose (RP2D).
- If 2/6 participants have DLT, 6 additional participants will be enrolled at starting dose level:
  - If a total of 2/12 participants treated at starting dose have DLT, starting dose will be the RP2D,
  - If a total of ≥3/12 participants have DLT, dose will be de-escalated to dose level minus 1 (DL-1).
- If  $\geq 3/6$  participants have DLT, dose will be de-escalated to DL-1.

An additional 6 participants may be enrolled at DL-1:

- If  $\leq 1/6$  participant has DLT, DL-1 will be the RP2D.
- If 2/6 participants have DLT, 6 additional participants will be enrolled at DL-1:
  - If a total of 2/12 participants treated at starting dose have DLT, DL-1 will be the RP2D,
  - If a total of  $\ge 3/6$  or  $\ge 3/12$  participants have DLT, an alternative dose/schedule might be considered from a safety viewpoint by the Sponsor.

Investigational medicinal product (IMP) initiation in each patient treated in Phase 1 is to be staggered by at least 3 days.

## 1.1.1.2 Dose limiting toxicity

Dose limiting toxicity (DLT) is defined in Section 4.1.1 in the protocol.

#### 1.1.1.3 Maximum tolerated dose and recommended Phase 2 dose

Any DLT observed during Cycle 1, and also overall safety including all the AEs occurring during treatment, unless due to disease progression or an obviously unrelated cause, will be taken into consideration by a Study Committee for the determination of the maximum tolerated dose (MTD) and RP2D for the isatuximab and atezolizumab combination.

The MTD is defined as the highest dose level at which no more than 1 out of 6 participants (starting dose or DL-1) or 2 out of 12 participants (starting dose) experience an IMP related DLT. The RP2D is defined as the dose selected for the Phase 2 portion.

## 1.1.2 Phase 2 (efficacy signal search with a 2-stage design in each cohort)

Phase 2 may include up to 6 cohorts: Cohorts A, B, C, and D-1 will be initiated in parallel, while other cohorts of the same tumor type will be open depending on results observed at the end of Stage 2 of the corresponding initial tumor type cohort.

- Cohort A: HCC, isatuximab and atezolizumab combination.
- Cohort B: SCCHN, isatuximab and atezolizumab combination.
- Cohort C: EOC, isatuximab and atezolizumab combination.
- Cohort D-1: GBM, isatuximab and atezolizumab combination.
- Possibly Cohort D-2: GBM, isatuximab monotherapy.
- Possibly Cohort E: isatuximab and atezolizumab combination in participants with one tumor type (HCC, SCCHN, EOC, or GBM), or isatuximab monotherapy (GBM only), without initial isatuximab weekly dosing.

12-Sep-2019 Version number: 1

A 2-stage design will be used in each cohort. Enrollment in Cohort D-2 may start only if clinical benefit is observed in Cohort D-1 at the end of Phase 2 Stage 2.

The participants treated at the RP2D of isatuximab and atezolizumab in combination during Phase 1 will be included in the efficacy analysis together with participants of the same tumor type in Phase 2 Stage 1. Based on the predefined number of objective responses in participants with SCCHN, HCC, EOC, or the predefined PFS-6 in participants with GBM, as well as any other relevant data observed within a treatment cohort in Phase 2 Stage 1, the study will proceed with Phase 2 Stage 2. After enrollment completion of Phase 2 Stage 1, if efficacy results do not warrant initiation of Stage 2, enrollment will be paused until sufficient results or analyses warrant initiation of Phase 2 Stage 2. In the case of inadequate efficacy for a cohort at interim analyses, the Sponsor will notify study sites regarding modification or termination of study procedures/scheduled activities for patients in that specific cohort.

For participants with GBM, if clinical benefit is observed in Cohort D-1 at the end of Phase 2 Stage 2, an isatuximab monotherapy cohort may be initiated (Cohort D-2). Participants with GBM will be enrolled into Cohort D-2, isatuximab monotherapy (Phase 2 Stage 1). The isatuximab single agent dose and schedule for Cohort D-2 will be determined based on results from Cohort D-1.

Based on the positive efficacy signal and the totality of data observed within a treatment cohort at end of Phase 2 Stage 2, the Sponsor may decide to further study in the same indication either isatuximab Q3W in combination with atezolizumab, or isatuximab Q3W as monotherapy in participants with GBM. This schedule without the initial weekly dosing may be more practical for participants and health care providers. Objectives and study design considerations for these cohorts are the same as those for other cohorts in the same tumor type, respectively.

#### 1.2 OBJECTIVES

#### 1.2.1 Primary objectives

## Phase 1:

• To characterize the safety and tolerability of isatuximab in combination with atezolizumab in participants with unresectable hepatocellular carcinoma (HCC), platinum-refractory recurrent/metastatic squamous cell carcinoma of the head and neck (SCCHN), platinum-resistant/refractory epithelial ovarian cancer (EOC), or recurrent glioblastoma multiforme (GBM), and to determine the recommended Phase 2 dose (RP2D).

#### Phase 2:

- To assess response rate (RR) of isatuximab in combination with atezolizumab in participants with HCC or SCCHN or EOC.
- To assess the progression free survival rate at 6 months (PFS-6) of isatuximab in combination with atezolizumab, or as a single agent in participants with GBM.

#### 1.2.2 Secondary objectives

- To evaluate the safety (in Phase 2) profile of isatuximab monotherapy (GBM only), or in combination with atezolizumab.
- To evaluate the immunogenicity of isatuximab and atezolizumab.
- To characterize the pharmacokinetic (PK) profile of isatuximab single agent (GBM only) and atezolizumab in combination with isatuximab.
- To assess overall efficacy of isatuximab in combination with atezolizumab, or single agent (GBM only).

#### 1.3 DETERMINATION OF SAMPLE SIZE

#### Phase 1

Approximately 6 (assuming 6 participants for the starting dose) to 24 (assuming 12 participants for the starting dose, and 12 participants for DL-1) DLT evaluable participants are expected to be enrolled. The actual sample size will vary depending on DLTs observed and the number of dose levels explored. Participants who are not evaluable for DLT assessment in Phase 1 may be replaced.

#### Phase 2

Phase 2 of the study is to evaluate initial anti-tumor activity based on tumor response using response evaluation criteria in solid tumors (RECIST) 1.1 criteria (1) for HCC, SCCHN and EOC, and response assessment in neuro-oncology (RANO) criteria (2) for GBM. The efficacy evaluation is based on 2-stage design with 85% power at 5% one-sided alpha level for each of the participant cohorts, respectively.

The assumption of RR, the required sample sizes, and the number of responders at each stage are provided in Table 2 for HCC, SCCHN and EOC:

Table 2 - Sample size calculation for HCC, SCCHN and EOC

| Indication | Н0 | H1 | Sample size | | | of responses<br>ect H0 |
|---|---|---|---|---|---|---|
| | | | Stage 1 | Final | Stage 1 | Final |
| HCC &<br>SCCHN | 15% | 30% | 26 | 59 | ≥5 (19.2%) | ≥14 (23.7%) |
| EOC | 20% | 40% | 17 | 37 | ≥4 (23.5%) | ≥12 (32.4%) |

Abbreviations: H0=null hypothesis; H1=alternative hypothesis; HCC=hepatocellular carcinoma; SCCHN=squamous cell carcinoma of the head and neck; EOC=epithelial ovarian cancer.

Note: Based on the number of objective responses and the totality of data observed within a treatment cohort in Phase 2 Stage 1, the Sponsor may decide to advance such a treatment cohort to Phase 2 Stage 2 after consulting with Study Committee.

12-Sep-2019 Version number: 1

The assumption of PFS-6, the required sample sizes, and PFS-6 at each stage are provided in Table 3 for GBM:

Table 3 - Sample size calculation for GBM

| Indication | dication H0 | H1 | Sample size | | Number (%) o<br>to reje | • |
|---|---|---|---|---|---|---|
| | | | Stage 1 | Final | Stage 1 | Final |
| GBM | 20% | 35% | 31 | 65 | >19.4% | >27.7% |

Abbreviations: H0=null hypothesis; H1=alternative hypothesis; GBM=glioblastoma multiforme.

Note: Based on the PFS-6 and the totality of data observed within a treatment cohort in Phase 2 Stage 1, the Sponsor may decide to advance such a treatment cohort to Phase 2 Stage 2 after consulting with Study Committee.

Participants who received the recommended dose regimen in Phase 1 will be also included in Phase 2 Stage 1 (eg, if 6 HCC participants were enrolled in Phase 1, only 20 HCC participants will be needed to complete the Phase 2 Stage 1 HCC cohort).

In Phase 2, approximately 285 participants are expected to be enrolled (assuming Cohort A, B, C, D-1, and D-2 complete 2 stages), including approximately 131 in Phase 2 Stage 1 and approximately 154 participants in Phase 2 Stage 2. The participants who are treated with RP2D in Phase 1 will be counted as Phase 2 participants.

If isatuximab Q3W in combination with atezolizumab or as monotherapy (GBM only) without the isatuximab QW for 3 weeks is to be tested in HCC, SCCHN, EOC, or GBM, 65 additional participants are expected to be enrolled. As a consequence, a total of up to 350 participants may be enrolled.

#### 1.4 STUDY PLAN

The complete study plan is presented in Section 1.2 of the protocol.

#### 1.5 MODIFICATIONS TO THE STATISTICAL SECTION OF THE PROTOCOL

The statistical section of the protocol was never changed in an amendment.

#### 1.6 STATISTICAL MODIFICATIONS MADE IN THE STATISTICAL ANALYSIS PLAN

Not applicable.

## 2 STATISTICAL AND ANALYTICAL PROCEDURES

Patients treated at the RP2D in Phase 1 will be included in the analysis with patients of the same tumor type in Phase 2. If the RP2D is the starting dose, all data from the patients in Phase 1 will be summarized together with the data from the patients of the same tumor type in Phase 2 except for the DLT analysis.

Data from HCC, SCCHN, EOC, and GBM cohorts (Cohorts A, B, C, D-1, and D-2) in Phase 2 will be analyzed and reported separately by cohort. Data from the cohort E will be summarized separately unless otherwise noted.

#### 2.1 ANALYSIS ENDPOINTS

## 2.1.1 Demographic and baseline characteristics

The baseline value is defined as the last assessment for this parameter before first administration of study treatments unless otherwise noted.

All baseline safety and efficacy parameters (apart from those listed below) will be presented along with summary statistics in the safety and efficacy sections (Section 2.4.5 and Section 2.4.6).

## Demographic characteristics

Demographic variables include race (American Indian or Alaska Native, Asian, Black or African American, Native Hawaiian or Other Pacific Islander, White, Not reported, Unknown), ethnicity (Hispanic or Latino, Not Hispanic or Latino, Not reported, Unknown), age in years, weight (kg), height (cm), eastern cooperative oncology group (ECOG) performance status (for patients with HCC or SCCHN or EOC) and Karnofsky performance status (for patients with GBM) at baseline.

#### Medical or surgical history

Medical or surgical history includes relevant history of previous or associated pathologies other than the tumor.

This information will be coded using the version of Medical Dictionary for Regulatory Activities (MedDRA) currently in effect at Sanofi at the time of database lock.

## Disease characteristics at diagnosis

The following disease characteristics at initial diagnosis will be described:

- Time from initial diagnosis to first study treatment administration (in years).
- Histology (diagnosis as collected in electronic case report form [eCRF]).
- Disease Location.

- Histopathology type (as collected in eCRF).
- Stage of the disease (as collected in eCRF, for patients with SCCHN and EOC).

## Disease characteristics at study entry - HCC

The following disease characteristics at study entry will be described:

- BCLC stage.
- Child-Pugh score.
- Progression on OR intolerance to other therapy.
- Extrahepatic metastases.
- Vascular invasion.

#### Disease characteristics at study entry - SCCHN

The following disease characteristics at study entry will be described:

- Tumor recurrence or PD within 6 months of last platinum-based therapy.
- HPV status.

## Disease characteristics at study entry - EOC

The following disease characteristics at study entry will be described:

- Disease resistant/refractory to platinum chemotherapy.
- BRCA1 status.
- BRCA2 status.

## Disease characteristics at study entry - GBM

The following disease characteristics at study entry will be described:

- IDH gene mutated.
- MGMT gene methyled.
- Surgeries undergone (complete resection, partial resection, biopsy only, other).

#### Prior anticancer therapies

Prior anti-cancer treatments are collected by regimen in the eCRF. The following variables will be summarized for each cohort (HCC, SCCHN, EOC, or GBM):

- Number of prior regimens (by category).
- Prior surgery related to disease: number (%) of patients with any prior surgery by type of procedure (Preferred Term).

In addition, for EOC cohort, prior PARP inhibitor will be summarized by category (0, 1 or >1).

Any technical details related to computation, dates, and imputation for missing dates are described in Section 2.5.

## 2.1.2 Prior or concomitant medications (other than anticancer therapies)

All medications will be coded using the World Health Organization-Drug Dictionary (WHO-DD), using the version currently in effect at Sanofi at the time of database lock.

- Prior medications are those the patient used prior to first study treatment administration.
   Prior medications can be discontinued before first dosing or can be ongoing during treatment phase.
- Concomitant medications are any treatments received by the patient concomitantly to the study treatment from first administration to the last administration + 30 days. A given medication can be classified both as a prior medication and as a concomitant medication.
- Post-treatment medications are those the patient took in the period running from the day after the last study treatment administration + 30 days up to the end of the study.

## Infusion associated reaction (IAR) medications

As defined in Section 6.6.4 of the study protocol, patients were to routinely receive premedications prior to isatuximab infusion to reduce the risk and severity of hypersensitivity reactions commonly associated with monoclonal antibodies. Premedications are defined in the protocol as non-investigational medicinal product(s). Premedications are reported on a specific eCRF page.

Any technical details related to computation, dates, imputation for missing dates are described in Section 2.5.

#### 2.1.3 Efficacy endpoints

#### 2.1.3.1 Primary efficacy endpoint(s)

The primary efficacy endpoint for the Phase 2 part of the study is RR for patients with HCC or SCCHN or EOC and is PFS-6 for patients with GBM.

For patients with HCC or SCCHN or EOC, the RR is defined as the proportion of patients with complete response and partial response as best overall response (BOR), assessed by investigators per RECIST 1.1 criteria, relative to the total number of patients in the analysis population. The confirmation of complete or partial response is required to determine BOR. BOR will be derived per RECIST 1.1 criteria using disease assessments performed from the first dose of treatment through the study excluding any assessments performed after the cut-off date or following the initiation of a further anticancer treatment. Clinical deterioration will not be considered as progression in the primary analysis of RR.

For patients with GBM, the PFS-6 is defined as the PFS rate at 6 months (assessed by Investigators per RANO criteria).

## 2.1.3.2 Secondary efficacy endpoint(s)

The secondary efficacy endpoints are:

- Tumor burden change: Tumor burden change is defined as the best percent-change from baseline in a sum of the diameters (longest for non-nodal lesion, short axis for nodal lesions) for all target lesions.
- Area under the curve (AUC) of percent-change from baseline in tumor burden is defined as the area under the percent-change from baseline versus time curve calculated using the trapezoidal method from the date of the first post-baseline assessment to the date of the last assessment.
- The time-adjusted AUC of percent-change from baseline in tumor burden is defined as AUC of percent-change from baseline in tumor burden divided by the duration of the assessment.
- Disease control rate (DCR): DCR is defined as the sum of the complete response (CR), partial response (PR) and stable disease (SD) rates. CR, PR, and SD are assessed by Investigator (per RECIST 1.1 criteria for HCC or SCCHN or EOC patients; per RANO criteria for GBM patients).
- Duration of response (DoR): DoR is defined as the time from the date of first response (PR or CR whichever is first) that is subsequently confirmed to the first date that recurrent or progressive disease progression is objectively documented, or the date of death, whichever occurs first. Disease progression refers to radiographic disease progression. The RECIST 1.1 criteria will be followed for assessment of radiographic disease progression in patients with HCC or SCCHN or EOC and the RANO criteria will be followed in patients with GBM. In the absence of disease progression or death before the analysis cut-off date or the date of initiation of a further anticancer treatment, the DoR will be censored at the date of the last valid response assessment not showing disease progression performed prior to initiation of a further anticancer treatment or the analysis cut-off date, whichever is earlier. DoR will not be calculated for patients who do not achieve a response.

Progression-free survival (PFS): PFS is defined as the time from first study treatment administration to the date of first documented radiographic progression (HCC, SCCHN, EOC per RECIST 1.1; GBM per RANO) or the date of death from any cause, whichever occurs first.

For patients who did not experience documented radiographic progression or death before the analysis cut-off date or the date of initiation of new anticancer treatment, PFS will be censored at the date of the last valid disease assessment not showing radiographic progression performed prior to initiation of a further anticancer treatment or the analysis cut-off date, whichever comes first. In addition, patient without PFS event (death or documented radiographic progression) and without any valid post-baseline disease assessments will be censored at the date of first treatment (Day 1).

• RR (GBM only): RR for GBM patients is defined as the proportion of patients with complete response and partial response as best overall response, assessed by Investigators using RANO criteria. The confirmation of complete or partial response is required to determine BOR. BOR will be derived per RANO criteria using disease assessments performed from the first dose of treatment through the study excluding any assessments performed after the cut-off date or following the initiation of a further anticancer treatment.

#### 2.1.3.3 Exploratory efficacy endpoint(s)

For patients with HCC, SCCHN, and EOC, the following endpoints will be summarized:

- RR, DCR, DoR, and PFS by modified Response Evaluation Criteria in Solid Tumors for immune-based therapies (iRECIST) (3). Definitions are similar to the ones in primary and secondary efficacy endpoints, except using iRECIST criteria instead of RECIST 1.1. Based on iRECIST, progressive disease should be confirmed on a second examination done at least 4 weeks apart to exclude pseudo progression. Once confirmed, the date of progression is the date of initial documented disease progression.
- Time to response (TTR): TTR is defined as the time from first study treatment administration to the first response (PR or CR whichever is first) that is subsequently confirmed (by RECIST 1.1 and iRECIST respectively).
- Time to progression (TTP): TTP is defined as the time from first study treatment administration to the date of first documented disease progression (by RECIST 1.1 and iRECIST respectively). Confirmation of progression is required by iRECIST. The date of progression is the date of initial documented disease progression.
- For patients who did not experience progression before the analysis cut-off date or the date of initiation of new anticancer treatment, TTP will be censored at the date of the last valid disease assessment not showing disease progression performed prior to initiation of a further anticancer treatment or the analysis cut-off date, whichever comes first. In addition, patient without disease progression and without any valid post-baseline disease assessments will be censored at the date of first treatment (Day 1).
- Overall survival (OS): OS is defined as the time from first study treatment administration to death from any cause. Patients without death prior to the analysis cut-off date will be censored at the last date the patient was known to be alive or the cut-off date, whichever comes first.

For patients with HCC, the following endpoint will also be summarized:

• Alpha-fetoprotein (AFP) reduction from baseline and relation with clinical response: % reduction and absolute reduction from baseline will be summarized for patients with clinical benefits (ie, patients with SD>6 months in the responder group) and others, respectively. Duration of SD is defined as the time from the date of first treatment to the date of first disease progression or death due to any cause, whichever occurs first.

For patients with EOC, the following endpoint will also be summarized:

• CA125 response by Gynaecologic Cancer Intergroup (GCIG) criteria and relation with clinical response. Patients should have a pre-treatment CA-125 of at least twice the ULN in order to be considered for CA-125 response. A CA-125 response would be obtained the moment the CA-125 is reduced by 50% and this should be confirmed with a consecutive CA-125 assessment not earlier than 28 days after the previous one, with however the date of the first 50% reduction to be the reference date for the CA-125 response. Patients are not evaluable by CA-125 if they have received mouse antibodies or if there has been medical and/or surgical interference with their peritoneum or pleura during the previous 28 days.

For patients with GBM, the following endpoints will be summarized:

- RR, DCR, DoR, and PFS by Immunotherapy Response Assessment in Neuro-Oncology (iRANO) (4). Definitions are similar to the ones in primary and secondary efficacy endpoints, except using iRANO criteria instead of RANO.
  - By iRANO, if it is  $\leq 6$  months after the initiation of immunotherapy, then a repeat scan is required to confirm radiographic progression. The minimum time interval for confirmation of progression is  $\geq 3$  months, and a new lesion dose not define PD.
  - By iRANO, if it is >6 months after the initiation of immunotherapy, then the confirmation of radiographic progression is not required, and a new lesion defines PD.
- OS-6: OS-6 is defined as the overall survival rate at 6 months.
- TTR and TTP (by RANO and iRANO). Definitions are similar to the ones for patients with HCC, SCCHN, and EOC, except using RANO and iRANO criteria.
- OS: Definition is same as OS for patients with HCC, SCCHN, and EOC.

#### 2.1.4 Safety endpoints

The safety analysis will be based on the reported adverse events (AEs) and other safety information, such as clinical laboratory data, vital signs, weight, electrocardiogram (ECG), Eastern Cooperative Oncology Group (ECOG) performance status (for patients with HCC or SCCHN or EOC) and Karnofsky performance status (for patients with GBM).

#### Observation period

The observation period starts from the time when the patient gives informed consent and is divided into 3 periods:

- The pre-treatment period is defined as the time informed consent is signed until the first dose of study treatments administration.
- The treatment-emergent adverse event (TEAE) period is defined as the time from the first dose of study treatments up to 30 days after last dose of study treatments.
- The post-treatment period is defined as the time starting from 31 days after the last dose of study treatments to the end of the study (as defined in the protocol).

## 2.1.4.1 Dose limiting toxicities (DLTs)

For the Phase 1 part dose limiting toxicities will be listed by patient using the DLT evaluable population.

#### 2.1.4.2 Adverse events variables

AEs (including serious adverse events [SAEs] and AEs of special interest [AESIs]) will be collected from the time of signed informed consent until the end of study.

## Adverse event observation period

- **Pre-treatment AEs** are defined as any adverse event reported during the pre-treatment period.
- **TEAEs** are adverse events that developed or worsened or became serious during the TEAE period.
- **Post-treatment AEs** are adverse events that developed or worsened or became serious during the post-treatment period.

All AEs (including SAEs and AESIs) will be graded according to NCI-CTCAE v4.03 and coded to a lower-level term, preferred term (PT), high-level term, high-level group term and associated primary system organ class (SOC) using the version of MedDRA currently in effect at Sanofi at the time of database lock.

#### Adverse events of special interest

Specific analyses will be performed for the following AEs:

- DLTs.
- Grade  $\geq 2$  acute IARs with isatuximab.
- Any grade IARs with atezolizumab.
- Grade ≥3 immune-related TEAEs.
- Any grade of the following TEAEs with atezolizumab: pneumonitis, colitis, endocrinopathies (diabetes mellitus, pancreatitis, adrenal insufficiency, hyperthyroidism, and hypophysitis), systemic lupus erythematosus, neurologic disorders (Guillain-Barré syndrome, myasthenic syndrome, myasthenia gravis, and meningoencephalitis), nephritis, ocular toxicities, myositis, myopathies, vasculitis, and autoimmune hemolytic anemia.
- Grade  $\geq 2$  cardiac disorders with atezolizumab.
- **Pregnancy** of a female patient entered in a study as well as pregnancy occurring in a female partner of a male patient entered in a study with IMP/non-investigational medicinal product (NIMP).
- **Symptomatic overdose** (serious or non-serious) with isatuximab/NIMP.

#### 2.1.4.3 Infusion associated reactions

Infusion associated reactions (IARs) typically occur within 24 hours from the start of each isatuximab/atezolizumab infusion.

Whenever possible, a diagnosis of the IAR (eg, Cytokine release syndrome, infusion related reaction, anaphylactic reaction, or any other teams chosen by the investigator) will be reported by the investigator in a specific AE page. In addition, symptoms of the IARs will be reported on a separate eCRF form.

IARs will be analyzed based on the investigator reported term collected in the specific AE pages.

#### 2.1.4.4 Deaths

The deaths will be summarized as follows:

- Deaths in TEAE period: includes all deaths occurring from the first IMP up to the end of treatment + 30 days.
- Deaths in post-treatment period: includes all deaths occurring after the end of TEAE period up to study closure.

## 2.1.4.5 Laboratory safety variables

Clinical laboratory data consists of blood and urine analysis including hematology, biochemistry and urinalysis. Clinical laboratory values will be converted into standard international units that will be used in all listings and tables.

Parameters measured on the day of the first study treatment infusion will be considered as part of the baseline measurements.

For laboratory safety variables, the treatment period is defined as the time from the first dose of study treatment (irrespective of treatment) administration to the last dose of study treatments + 30 days.

Blood and urine samples for clinical laboratories parameters will be taken as defined in the study flow charts and as clinically indicated. The laboratory parameters will be classified as follows:

- Hematology
  - **Hemoglobin and coagulation**: hemoglobin, hematocrit, red blood cell (RBC) count, platelet counts, prothrombin time or international normalized ratio (INR) and activated partial thromboplastin time (PTT).
  - White blood cells (WBCs): leukocytes, neutrophils, lymphocytes, monocytes, basophils, eosinophils.
- Biochemistry
  - **Metabolism**: fasting glucose, total protein,

- **Electrolytes**: sodium, potassium, chloride, calcium, albumin, magnesium, phosphate, bicarbonate/carbon dioxide,
- **Renal function**: uric acid, serum creatinine, estimated creatinine clearance by modified diet in renal disease (MDRD) formula, urea or blood urea nitrogen (BUN),
- **Liver parameters**: alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase, total and direct bilirubin, lactate dehydrogenase (LDH).
- **Hormonal**: thyroid stimulating hormone (TSH) and free T4.
- Urinalysis
  - Quantitative or semi-quantitative urinalysis: RBC, protein, glucose, pH, leukocytes.

## 2.1.4.6 Vital signs variables

Vital signs include: weight, temperature, pulse rate, systolic and diastolic blood pressure, and respiratory rate. Oxygen saturation is assessed for patients with SCCHN only.

Weight is required at Screening, prior to starting infusion and at the EOTvisit. Temperature, pulse rate, respiratory rate, and blood pressure will be performed at screening, at Cycle 1 Day 1, Day 8 and Day 15, and Cycle N Day 1 - just before starting infusion of IMPs, during infusion, and at the end of infusion, at EOT visit, and at post treatment follow-up visits at 60 and 90 days after last treatment.

Thus, parameters measured pre-infusion on the day of the first study treatment infusion will be considered as part of the baseline measurements.

For a given parameter, a patient (respectively a cycle) will be considered as evaluable if at least one measure of this parameter is available during the on-treatment period.

## 2.1.4.7 Electrocardiogram variables

12-lead ECG assessments will be described as normal or abnormal.

#### 2.1.4.8 Clinical safety laboratory assessments

All protocol-required laboratory assessments, as defined in Section 10.3 of the protocol, will be performed and to the Schedule of Activities for the timing and frequency.

The Investigator must review the laboratory report, document this review, and record any clinically relevant changes occurring during the study in the AE section of the eCRF. Remaining laboratory tests are reported in eCRF pages for Hematology and Biochemistry.

All laboratory tests with values considered clinically significantly abnormal during participation in the study or after the last dose of study intervention should be repeated until the values return to normal or baseline or are no longer considered clinically significant by the Investigator or Medical Monitor. If such values do not return to normal/baseline within a period of time judged reasonable by the Investigator, the etiology should be identified.

#### 2.1.4.9 Immunogenicity variables

Anti-drug antibodies (ADA) against isatuximab and atezolizumab will be collected according to the pharmacokinetics/pharmacodynamics (PK/PD) flowcharts in Section 1.3 of the protocol.

#### ADA attributes

**Pre-existing ADA** is defined as ADA reactive with the biotherapeutic present in subjects before treatment (or before initiation of the clinical study).

**Treatment boosted ADA** is defined as pre-existing ADAs that were boosted to a higher level following administration of biotherapeutic (ie, any time after the initial drug administration) the ADA titer is significantly higher than the baseline titer. A low serial dilution schema (2-fold or 3 fold) should be applied during titration. A difference in titer values of two titer steps between treatment or follow-up sample and its baseline sample is considered significant. For examples, at least a 4-fold increase in titers for 2- fold serial dilution schema (or 9-fold increase in titers for 3- fold serial dilution schema). If no titer could be determined for a positive sample, the titer will be reported as the minimal required dilution of the assay.

**Treatment-induced ADA** is defined as ADAs developed de novo (seroconversion) following administration of the biotherapeutic (ie, formation of ADAs any time after the initial drug administration in a subject without pre-existing ADAs). If the baseline ADA sample is missing or non-reportable and at least one reportable ADA sample is available during the treatment (including follow-up period) the baseline sample will be considered as "negative" for data analysis. This is considered being a conservative approach for ADA assessment.

## Subject status

Among evaluable population for immunogenicity (described in Section 2.3.5), following patient status will be defined:

- **ADA-positive** subject: A subject with at least one treatment induced or treatment boosted ADA-positive sample at any time during the treatment or follow-up observation period.
- **ADA-negative** subject: Subject without any treatment induced or treatment boosted ADA-positive sample during the treatment or follow-up observation period.
- **ADA-inconclusive** subject: A subject who cannot irrefutably be classified as ADA negative (eg, all post baseline samples inconclusive).

## Overview of the ADA response

Two main categories can be reported for the epidemiology of an ADA immune response: ADA prevalence and ADA incidence:

• ADA prevalence defines the proportion of all subjects tested positive for ADAs (including preexisting antibodies, treatment boosted ADAs and treatment induced ADAs) at any point in time.

• In contrast the term **ADA incidence** only defines the proportion of subjects found to either have seroconverted (treatment induced ADAs) or boosted their pre-existing ADA response during the study. Only evaluable subjects (described in Section 2.3.5) are considered for computing ADA incidence.

## Kinetics of the immune response

- Onset of ADA: refers to the time period between the initial drug administration and the first instance of treatment induced ADAs. The use of real-elapsed days should be used for the calculations. The "median time to ADA development" and the quartiles Q1 and Q3 should be reported.
- **Duration of ADA:** ADA duration will be calculated as the date of last treatment induced ADA sample minus date of first treatment induced or treatment boosted ADA sample +1; ADA duration will be calculated only for patients with at least two ADA positive samples. Median duration of an induced ADA response and the quartiles Q1 and Q3 should be reported.
- Transient ADA response is defined by:
  - Treatment induced ADA detected only at one sampling time point during the treatment or follow-up observation period (excluding the last sampling time point), OR
  - Treatment induced ADA detected at two or more sampling time points during the treatment (including follow-up period if any), where the first and last ADA-positive samples (irrespective of any negative samples in between) are separated by a period less than 16 weeks, and the patient's last sampling time point is ADA negative.
- **Persistent ADA response** is defined by:
  - Treatment induced ADA detected at two or more sampling time points during the treatment (including follow-up period if any), where the first and last ADA-positive samples are separated by at least 16 weeks (irrespective of any negative samples in between).
- Indeterminate ADA is defined by:
  - Treatment induced ADA detected only at the last sampling time point, OR
  - The last two samples being ADA-positive and separated by a period of less than 16 weeks.

Treatment-boosted ADAs are excluded from the analysis of ADA kinetics.

#### 2.1.5 Pharmacokinetic variables

PK analysis will be done separately for isatuximab and atezolizumab.

The PK sampling times for isatuximab and atezolizumab were provided in the PK/PD flowchart in Section 1.3 of the protocol.

• For isatuximab only: the following PK parameters (listed in Table 4) will be calculated with PKDMS software (Pharsight) V3.0, using non-compartmental method from isatuximab concentrations after the first administration on Cycle 1. The parameters will include, but may not be limited to the following:

Table 4 - List of pharmacokinetic parameters and definitions

| Parameters | Analyte | | Definition |
|---|---|---|---|
| | Atezolizumab | Isatuximab | - |
| Ceoi | Х | Х | Concentration observed at the end of intravenous (IV) infusion |
| Cmax | Х | Χ | Maximum concentration observed |
| tmax | Χ | Χ | Time to reach Cmax |
| Clast | Х | Χ | Last concentration observed above the lower limit of quantification |
| tlast | Х | Χ | Time of Clast |
| AUC0-7d | Х | | Area under the concentration versus time curve calculated using the trapezoidal method over the dosing interval (21 days) |

• For isatuximab and atezolizumab: C<sub>trough</sub> defined as sample collected just before treatment administration and C<sub>eoi</sub> will be measured over the study period.

In addition, populations PK approaches may be used for both compounds and PK estimates may be used to conduct exploratory exposure-response analyses for safety and efficacy and PK/PD analyses for relevant biomarkers. If done, the data generated will be reported in stand-alone report(s).

## 2.1.6 Biomarker endpoints

#### 2.1.6.1 Microsatellite instability

Microsatellite instability will be analyzed on tumor samples collected at screening or baseline:

• Results will be of the form of MSI-H (ie, high microsatellite instability) or no-MSI-H (ie, low microsatellite instability or microsatellite stable).

#### 2.1.6.2 PD-L1 expression singleplex IHC

PD-L1 expression on tumor and immune cells will be assessed using tumor tissue (freshly collected tumor biopsy or archival tissue) biopsy at Screening/Baseline and (unless clinically unfeasible) at C2D1.

## 2.1.6.3 Cluster of differentiation 38 (CD38) expression singleplex IHC

CD38 expression on tumor and immune cells will be assessed using tumor tissue (freshly collected tumor biopsy or archival tissue) biopsy at Screening/Baseline and (unless clinically unfeasible) at C2D1.

# 2.1.6.4 Immune cell subpopulation tumor infiltration and markers co-expression multiplex immunofluorescence

Immune cell subpopulation tumor infiltration and markers co-expression on different cell sub-populations will be assessed on tumor tissue (freshly collected tumor biopsy or archival tissue) biopsy at Screening/Baseline and (unless clinically unfeasible) at C2D1. Cell sub-populations will be determined by multiplex Immunofluorescence based on the expression of 12 different cell markers. The results will be provided per region of interest (ROI) and the number of cell sub-populations will be provided for 3 regions (total, within tumor, outside tumor).

Per cell sub-population, an average of the results provided per ROI will be calculated for the totality of tumor tissue.

# 2.1.7 Further therapy after discontinuation of investigational medicinal product administration during the study

Further therapies after discontinuation of study treatment will be collected on a specific eCRF page. The following information will be collected: drug/medication (brand or generic name), start date and end date (if available)/ongoing (otherwise).

#### 2.2 DISPOSITION OF PATIENTS

Patient disposition will be summarized by cohort based on the analysis population defined in Section 2.3.

Screened patients are defined as any patients who signed the study informed consent.

Enrolled patients are screened patients who are planned to receive the study treatment, ie, for whom the investigator ticked "Yes" to the question "Will the patient continue into the study?" at the end of the screening period.

For patient study status, the total number of patients for each of the following categories will be presented in the clinical study report using a flow-chart diagram or a summary table:

- Screened patients.
- Enrolled patients.
- Enrolled and not treated patients.
- Enrolled and treated patients.
- Patients still on treatment.
- Patients completed treatment.
- Patients who discontinued the study treatments period and reasons for permanent discontinuation.

12-Sep-2019 Version number: 1

The number and percentage of patients in analysis population (defined in Section 2.3) will be provided in a summary table.

A summary of the reasons for definitive and premature treatment discontinuation for either treatment will be provided. Definitive treatment discontinuation is defined as the discontinuation of all the study treatments. Premature treatment discontinuation (only for cohorts with the combination therapy) is defined as the discontinuation of one of the study treatments but the other one continued. Listing of the reasons for treatment discontinuation will be provided.

The number (%) of patients treated by country and center will be summarized using the all-treated population (defined in Section 2.3).

All critical or major deviations potentially impacting efficacy and safety analyses will be summarized by cohort separately. Critical or major protocol deviations will be listed.

#### 2.2.1 Randomization and drug dispensing irregularities

This is an open-label, non-randomized study; therefore, randomization and dispensing irregularities are not applicable.

#### 2.3 ANALYSIS POPULATIONS

#### 2.3.1 All-treated population

For both Phase 1 and Phase 2 parts of the study, the all-treated population will include all patients who signed the study informed consent and received at least 1 dose (even incomplete) of the study treatments, either isatuximab or atezolizumab.

This population is the primary population for the analyses of efficacy and safety parameters except for DLT evaluation. All analyses using this population will be based on the dose level actually received in the first cycle.

#### 2.3.2 DLT-evaluable population

The DLT evaluable population is defined as patients in the Phase 1 part receiving the planned doses of isatuximab and atezolizumab during Cycle 1, and who completed the DLT observation period after the first IMP administration as per Section 4.1.1 from protocol, unless they discontinue the study treatment(s) due to DLT. The dose recommended for Phase 2 will be determined on the DLT evaluable population.

#### 2.3.3 Pharmacokinetic population

The PK population will be defined independently for isatuximab and atezolizumab, and include patients from the all treated population who received at least one dose of the drug even if incomplete with at least one reportable concentration after the study drug administration (whatever the cycle and even if dosing is incomplete).

## 2.3.4 Biomarker Population

The biomarker population will include all treated patients who submitted at least one baseline biomarker sample.

## 2.3.5 Immunogenicity population

The immunogenicity population will be defined independently for isatuximab and atezolizumab, and include subjects from the all treated population who received at least one dose of the drug even if incomplete with at least one sample, taken post-baseline after drug administration during the treatment or follow-up observation period, with a reportable result (positive, negative or inconclusive).

#### 2.3.6 Response evaluable population

The response evaluable population will include all patients in the all-treated population who fulfilled all inclusion and exclusion criteria with an evaluable baseline assessment and at least one evaluable post-baseline disease assessment during the treatment period.

#### 2.4 STATISTICAL METHODS

Continuous data will be summarized using number of available data, mean, standard deviation, median, minimum and maximum for each dose level (if applicable). Categorical and ordinal data will be summarized using number and percentage of patients.

Data listings will be provided separately by cohort and sorted by patient number, unless otherwise specified.

#### 2.4.1 Demographics and baseline characteristics

Demographics and baseline characteristics will be summarized on the all-treated population. Parameters described in Section 2.1.1 will be summarized using descriptive statistics.

The medical and surgical history will be summarized according to the SOC and PT (SOC will be sorted according to the internationally agreed order and PT by overall decreasing frequency).

Disease characteristics at diagnosis and at study entry will be described.

## 2.4.2 Prior or concomitant medications (other than anticancer therapies)

The prior, concomitant and post medications will be presented for the all-treated population. The anti-cancer therapy will be presented separately.

Medications will be summarized according to the WHO-DD dictionary, considering the first digit of the anatomic therapeutic category (ATC) class and the first 3 digits of the ATC class (therapeutic category). All ATC codes corresponding to a medication will be summarized, and the

12-Sep-2019 Version number: 1

patients will be counted once in each ATC category (anatomic or therapeutic) linked to the medication. Therefore the patients may be counted several times for the same medication.

The tables for medications (prior, concomitant and post-treatment) will be sorted by decreasing frequency of ATC followed by all other therapeutic classes based on the overall incidence. In case of equal frequency regarding ATCs, alphabetical order will be used.

#### IAR medications

Number (%) of patients with IAR medications as defined in Section 2.1.2 will be provided.

## 2.4.3 Anticancer therapies

Prior anti-cancer treatments will be summarized for the all-treated population. Number (%) of patients with the anti-cancer treatments described in Section 2.1.1 will be summarized.

## 2.4.4 Extent of investigational medicinal product exposure and compliance

The extent of study treatment exposure will be assessed and summarized on the all-treated population.

## 2.4.4.1 Extent of investigational medicinal product exposure

The overall extent of exposure will be assessed as:

- Overall number of cycles started.
- Duration of overall exposure (weeks): defined as (last day of last cycle first day of first cycle)/7. The first day of first cycle is defined as the date of the first dose of study treatments. The last day of last cycle is defined as the later date among the following:
  - Date of the last dose of isatuximab + 7 days if the last cycle is a QW cycle or date of the last dose of isatuximab + 21 days if the last cycle is a Q3W,
  - Date of the last dose of atezolizumab + 21 days.

Total number of cycles started, number of cycles started by patient as a continuous variable and by category (ie, number [%] of patients receiving at least 1 cycle, at least 2 cycles, etc), duration of overall exposure will be summarized using descriptive statistics.

To describe overall dose modification, the cycle delay will be summarized. A cycle is considered as delayed if the start date of cycle - 21 - the start date of the previous cycle is >3 days. The cycle start date is defined as the earlier date of isatuximab or atezolizumab administration within a cycle. Cycle delay is not defined for the first cycle.

Cycle delay will be summarized at both the patient and cycle levels as follows:

- Patient level:
  - Number of patients treated,
  - Number (%) of treated patients with at least 1 cycle delayed,
    - Number (%) of treated patients with a cycle delayed between 4 and 7 days,
    - Number (%) of treated patients with a cycle delayed between 8 and 14 days,
    - Number (%) of treated patients with a cycle delayed more than 14 days.
- Cycle level:
  - Number of cycles started,
  - Number (%) of cycles delayed,
    - Number (%) of cycles delayed between 4 and 7 days,
    - Number (%) of cycles delayed between 8 and 14 days,
    - Number (%) of cycles delayed more than 14 days.

## 2.4.4.2 Isatuximab exposure

The isatuximab exposure will be summarized as follows:

- Total number of cycles started.
- Number of cycles started by patient as a continuous variable and by category.
- Duration of isatuximab exposure (weeks) is defined as:
  - (Date of the last dose of isatuximab + 7 days date of the first dose of isatuximab)/7 if the last cycle is a QW cycle,
  - (Date of the last dose of isatuximab + 21 days date of the first dose of isatuximab)/7 if the last cycle is a Q3W cycle.
- Actual dose (mg/kg): is defined as the actual dose (mg) administered divided by the body weight at the time.
- Cumulative dose (mg/kg): the cumulative dose is the sum of all actual doses (mg/kg) of isatuximab given from the first to the last administration.
- Actual dose intensity (ADI, mg/kg/week): is defined as the cumulative dose (mg/kg) divided by the duration of isatuximab exposure (weeks).
- Relative dose intensity (RDI, %):  $100 \times \frac{\text{ADI}(\text{mg/kg/week})}{\text{Planned Dose Intensity (mg/kg/week)}}$ .

Planned dose intensity (mg/kg/week) corresponds to the planned dose (mg/kg) multiplied by the theoretical total number of doses during the started cycles (3 for QW cycle and 1 for Q3W cycle) and divided by the theoretical cycle duration (weeks), ie, 3 weeks per cycle started.

The total number of cycles started, number of cycles started by patients as a continuous variable and by category (ie, number [%] of patients receiving at least 1 cycle, at least 2 cycles, etc), duration of isatuximab exposure, cumulative dose, ADI and RDI will be summarized by descriptive statistics.

The following variables will be derived to describe dose delay and modification:

- Dose delay within Cycle 1: a dose is deemed as delayed within Cycle 1 if the actual start date of the infusion is ≥2 days beyond the theoretical day of treatment for weekly dose. Dose delay does not apply to the first infusion of Cycle 1.
- Infusion interruption: an infusion is considered to be interrupted (as collected on eCRF) if the isatuximab administration is stopped during an infusion before it is completed regardless of whether it is further restarted or not.
- Dose omission: a dose is considered omitted if the dose is not administered for the scheduled visit and there are dose(s) administered afterwards.

Dose delay and modification will be summarized at the patient and infusion levels as follows:

- Patient level:
  - Number (%) of patients with at least 1 dose delay within cycle,
  - Number (%) of patients with at least 1 dose omission,
  - Number (%) of patients with at least 1 infusion interrupted,
    - Number (%) of patients with at least 1 infusion interrupted and re-started,
    - Number (%) of patients with at least 1 infusion interrupted and not re-started.
- Infusion level:
  - Number of isatuximab infusions,
  - Number (%) of infusions interrupted,
    - Number (%) of infusions interrupted and re-started,
    - Number (%) of infusions interrupted and not re-started,
  - Number (%) of infusions interrupted more than once,
  - Number (%) of infusions interrupted at 1st infusion, 2nd infusion, subsequent infusions.
  - Time from infusion start to first interruption in minutes summarized as a continuous variable and by category (<5 minutes, 5-10 minutes, etc).

#### 2.4.4.3 Atezolizumab exposure

The atezolizumab exposure will be summarized as follows:

- Total number of cycles started.
- Number of cycles started by patient as a continuous variable and by category.
- Duration of atezolizumab exposure (weeks) is defined as (Date of the last dose of atezolizumab + 21 days Date of the first dose of atezolizumab)/7.

- Actual dose (mg): is defined as actual dose administered.
- Cumulative dose (mg): the cumulative dose is the sum of all actual atezolizumab doses.
- ADI (mg/week): is defined the cumulative dose (mg) divided by the duration of atezolizumab exposure (weeks).
- RDI (%): 100× ADI (mg/week) Planned Dose Intensity (mg/week), where the planned dose intensity (mg/week) is 400 mg/week for Q3W schedule.

The total number of cycles started, number of cycles started by patients as a continuous variable and by category (ie, number [%] of patients receiving at least 1 cycle, at least 2 cycles, etc), duration of atezolizumab exposure, cumulative dose, ADI and RDI will be summarized by descriptive statistics.

The following variables will be derived to describe dose delay and modification:

- Infusion interruption: An infusion will be considered to be interrupted (as collected on eCRF) if the atezolizumab administration is stopped during an infusion before it is completed regardless of whether it is further restarted or not.
- Dose omission: a dose is considered omitted if the dose is not administered for the scheduled visit and there are positive dose(s) afterwards.

Dose delay and modification will be summarized at the patient and infusion levels as follows:

- Patient level:
  - Number (%) of patients with at least 1 dose omission,
  - Number (%) of patients with at least 1 infusion interrupted,
    - Number (%) of patients with at least 1 infusion interrupted and re-started,
    - Number (%) of patients with at least 1 infusion interrupted and not re-started.
- Infusion level:
  - Number of atezolizumab infusions,
  - Number (%) of infusions interrupted,
    - Number (%) of infusions interrupted and re-started,
    - Number (%) of infusions interrupted and not re-started,
  - Number (%) of infusions interrupted more than once,
  - Number (%) of infusions interrupted at 1st infusion, 2nd infusion, subsequent infusions,
  - Time from infusion start to first interruption in minutes summarized as a continuous variable and by category (<5 minutes, 5-10 minutes, etc).

## 2.4.5 Analyses of efficacy endpoints

All efficacy analysis will be performed using the all-treated population. In addition, efficacy analysis will be performed using the response evaluable population.

For each cohort, the analysis cut-off date for the primary analysis (RR for HCC, SCCHN, and EOC; PFS-6 for GBM) will be 6 months after the last participant's first treatment in the cohort.

The analysis cut-off date for secondary efficacy endpoints including DoR and PFS will be 12 months after the last participant's first treatment in the cohort. The primary analysis of RR in the cohort for HCC, SCCHN, and EOC, and of PFS-6 in the cohort for GMB will be updated. In case of inadequate efficacy for a cohort at interim analyses, the Sponsor may decide not to update primary nor perform secondary analyses for that cohort.

## 2.4.5.1 Analysis of primary efficacy endpoint(s)

For HCC, SCCHN and EOC, RR will be summarized with descriptive statistics. A 90% 2-sided confidence interval will be computed using Clopper-Pearson method. BOR will be summarized descriptively.

For GBM, PFS-6 will be summarized using Kaplan-Meier method.

## 2.4.5.2 Analyses of secondary efficacy endpoints

The analyses of secondary efficacy endpoints include:

- Tumor burden change: the best percent-change from baseline in tumor burden will be summarized and presented graphically for patients with measurable disease at baseline. In addition, a summary of the AUC and the time-adjusted AUC of percent-change from baseline in tumor burden will also be provided as an exploratory analysis.
- DCR: DCR (complete response + partial response + stable disease) will be summarized with descriptive statistics.
- DoR: Kaplan-Meier estimates such as median and Kaplan-Meier curves will be provided for patients who achieved a response (PR or CR).
- PFS: the PFS will be analyzed using the Kaplan-Meier method. The Kaplan-Meier estimates of the 25th, 50th and 75th percentiles and the 95% confidence intervals of median will also be computed. The Kaplan-Meier curves will be plotted. In addition, PFS at 6 months will also be provided.
- RR (GBM only): RR for GBM patients will be summarized with descriptive statistics.

#### 2.4.5.3 Analyses of exploratory efficacy endpoints

RR and DCR by iRECIST for patients with HCC, SCCHN and EOC, as well as by iRANO for GBM patients, will be summarized with descriptive statistics.

For patients with HCC, SCCHN and EOC, Kaplan-Meier method will be used to analyze DoR and PFS by iRECIST, TTR and TTP by RECIST 1.1 and iRECIST respectively, and OS.

For patients with GBM, Kaplan-Meier method will be used to analyze DoR and PFS by iRANO, TTR and TTP by RANO and iRANO respectively, OS-6, and OS.

In addition, AFP reduction from baseline for HCC patients and CA125 response for EOC patients will be summarized with descriptive statistics.

#### 2.4.5.4 Multiplicity issues

Not applicable.

## 2.4.6 Analyses of safety data

The all-treated population will be used for all safety analyses except for the DLT analysis in Phase 1, which will be performed based on the DLT-evaluable population.

## 2.4.6.1 Analyses of DLTs (Phase 1 only)

The DLTs will be listed by patient using the DLT-evaluable population in Phase 1.

#### 2.4.6.2 Analyses of adverse events

The primary focus of adverse event reporting will be on treatment-emergent adverse events. Pre-treatment and post-treatment adverse events will be described separately.

If an AE date of onset (occurrence, worsening, or becoming serious) is incomplete, an imputation algorithm will be used to classify the AE as pretreatment, treatment-emergent, or post-treatment. The algorithm for imputing date of onset will be conservative and will classify an AE as treatment emergent unless there is definitive information to determine it is pretreatment or post-treatment. Details on classification of adverse events with missing or partial onset dates are provided in Section 2.5.3.

Regarding treatment discontinuation, following definitions will be used:

- **Premature** treatment discontinuation is defined when 1 of the IMPs is permanently discontinued, subjects will continue receiving the other IMP until study treatment permanent discontinuation.
- **Definitive** treatment discontinuation is defined as the discontinuation of all the study drugs.

The severity grade will be taken into account in the summary. For patients with multiple occurrences of the same AE, the maximum (worst) severity grade by period of observation will be used. Summaries will be provided for all grades and for Grade  $\geq 3$  (including Grade 5). Missing grades handling is provided in Section 2.5.3.

Sorting within tables should ensure the same presentation for the set of all AEs for each observation period (pre-treatment, treatment-emergent and post-treatment). For that purpose, tables of all TEAEs by SOC and PT will be sorted by the internationally agreed SOC order and decreasing frequency of PTs within SOCs. This order will define the presentation order for all other tables unless otherwise specified.

## Overall summary of TEAEs

An overall summary of TEAEs will be provided. The number (%) of patients who experience any of the following will be provided:

- TEAE.
- TEAE of Grade  $\geq 3$ .
- TEAE of Grade 5.
- Serious TEAE.
- Treatment-related TEAEs (any grade).
- Treatment-related TEAEs of Grade >3.
- Serious treatment-related TEAEs.
- TEAE leading to definitive study treatment discontinuation.
- TEAE leading to premature discontinuation of isatuximab.
- TEAE leading to premature discontinuation of atezolizumab.
- AESI.
- AESI of Grade  $\geq 3$ .

#### Analysis of all TEAEs

The number (%) of patients experiencing TEAEs by primary SOC and PT will be summarized by grade (all grades and Grade ≥3). Similar tables will be presented for treatment-related TEAEs, serious TEAEs, and TEAEs leading to definitive/premature discontinuation.

TEAEs with an incidence  $\geq$ 5% will be summarized by PT for all grades and Grade  $\geq$ 3.

Listings of serious TEAEs, TEAEs leading to definitive or premature treatment discontinuation will be provided.

## Infusion associated reactions (IARs)

IAR analysis will include all adverse events regardless of relationship to isatuximab, atezolizumab or NIMP. The IARs will be summarized as follow:

- Number (%) of patients experiencing IARs according to investigator reported AEs presented by primary SOC and PT will be summarized by grade.
- Description of the IAR diagnoses (using the diagnosis reported and excluding symptoms).
  - Number (%) of patients action taken,
  - Number (%) of patients with only  $1, \ge 1, \ge 2, \ge 3, \ge 4$  and  $\ge 5$  episodes,
  - Number (%) of patients with first occurrence of IAR at the first infusion and subsequent infusions,
  - Number (%) of patients with IAR at the first and subsequent infusions,
  - Number (%) of patients with at least two episodes of IRs at the same infusion,
  - Day of onset from infusion,
  - Duration (in days).
- Number of patients with symptoms of IARs (as reported by investigator) by SOC and PT.

## Analysis of adverse events of special interest

A listing of patients with at least one AESI described in Section 2.1.4.2 will be provided.

#### Analysis of pre-treatment and post-treatment adverse events

The following analysis will be provided by grade (all grades and Grade  $\geq 3$ ).

- All pre-treatment AEs by primary SOC and PT, showing the number (%) of patients with at least 1 pre-treatment AE, sorted by the internationally agreed SOC order and decreasing incidence of PTs within each SOC.
- All post-treatment AEs by primary SOC and PT, showing the number (%) of patients with at least 1 post-treatment AE, sorted by the internationally agreed SOC order and decreasing incidence of PTs within each SOC.

#### 2.4.6.3 Deaths

The following summaries of deaths will be generated:

- Number (%) of patients who died by study period (on-treatment, post-treatment) and reasons for death (disease progression, AE, other).
- TEAEs with fatal outcome (on the AE eCRF page as reported by the Investigator), TEAEs that started as non-fatal during treatment period but became fatal during post-treatment period, and TEAEs with fatal outcome during the post-treatment period summarized by SOC and PT.

## 2.4.6.4 Analyses of laboratory variables

Each laboratory test result will be graded by CTCAE criteria (version 4.03), when applicable. For hematological parameters and for some biochemistry parameters, Sanofi sponsor generic normal ranges will be used for the grading of laboratory abnormalities (see list of parameters in Table 7 and Table 8). For other biochemistry parameters (eg, for hepatic parameters), grading will be derived using the local laboratory normal ranges.

The number (%) of patients with abnormal laboratory tests at baseline and during the on-treatment period will be presented by all grades and each grade. For patients with multiple occurrences of the same laboratory variable during the on-treatment period, the maximum grade (worst) per patient will be used.

The denominator used for percentage calculation is the number of patients with at least 1 evaluation of the laboratory test during the considered observation period.

When appropriate, the summary table will present the frequency of patients with any grade of abnormal laboratory tests and with Grade 3-4 abnormal laboratory tests.

## 2.4.6.5 Analyses of vital sign variables

The incidence of vital signs potentially clinically significant abnormality (PCSA) (Table 5) any time during the on-treatment period will be summarized by treatment group irrespective of the baseline level and/or according to the following baseline status categories:

- Normal/missing.
- Abnormal according to PCSA criterion or criteria.

Table 5 - Potentially clinically significant abnormalities criteria for vital signs

| Parameter | PCSA |
|---|---|
| HR | ≤50 bpm and decrease from baseline ≥20 bpm ≥120 bpm and increase from baseline≥20 bpm |
| SBP | ≤95 mmHg and decrease from baseline ≥20mmHg<br>≥160 mmHg and increase from baseline ≥20 mmHg |
| DBP | ≤45 mmHg and decrease from baseline ≥10 mmHg<br>≥110 mmHg and increase from baseline ≥10 mmHg |
| Weight | ≥5% increase from baseline<br>≥5% decrease from baseline |

Temperature and respiratory rate will be summarized at baseline and end of treatment. A listing of patients with at least one PCSA will be provided.

## 2.4.6.6 Analyses of electrocardiogram variables

A listing of patients with ECG results will be provided.

#### 2.4.6.7 Analysis of Immunogenicity

Immunogenicity analysis will be done separately for isatuximab and atezolizumab.

Number of evaluable patients, number (%) of pre-existing ADA and negative patients at baseline, number (%) of boosted and induced patients (either transient, persistent or indeterminate) will be reported, along with descriptive statistics of titer, by cohort and possibly overall. Prevalence and incidence will also be presented.

In addition, for positive ADA patients, time to onset, duration of ADA response, and the characterization of the immune response (transient, persistent, indeterminate) will be provided.

An individual data listing with ADA samples status (positive, negative or inconclusive), the titer if applicable, date of first/last dose, duration of exposure, study period, cycle/day, time point and date/time of sampling along with Ctrough value of the drug will be provided for all patients.

The impact on safety and efficacy endpoints may be further explored by graphical methods or descriptively, depending on the ADA prevalence.

#### 2.4.7 Analyses of pharmacokinetic variables

# 2.4.7.1 Cycle 1 non-compartmental analysis of isatuximab: following the 1<sup>st</sup> administration

Following the first administration, individual concentrations and PK parameters of drug will be listed and summarized by descriptive statistics (such as the number of observations, arithmetic and geometric mean, median, SD, SEM, CV%, minimum, and maximum) by cohort and overall. Individual and mean concentration profiles over time will be plotted by cohort and overall under the responsibility of Sanofi, Pharmacokinetic, Dynamic and Metabolism (PKDM), Translational Medicine and Early Development (TMED) department.

#### 2.4.7.2 Over treatment concentrations: Ctrough and Ceoi of isatuximab and atezolizumab

Ctrough defined as a sample collected before dosing, in a time window of 6 to 8 days after the previous infusion for the QW administration and in a time window of 18 to 24 days after the previous infusion for the Q3W administration (always before administration) will be included in the descriptive analysis irrespectively of interruption of infusion. However Ctrough drawn outside time collection window described in the protocol PK flowchart or collected after a dose deviation higher than  $\pm 50\%$  from intended dose will be excluded from the analyses.

Ceoi (only for isatuximab) collected after a dose deviation higher than  $\pm 50\%$  from intended dose will be excluded from the analyses.
12-Sep-2019 Version number: 1

Individual Ctrough and Ceoi (only for isatuximab) will be listed and summarized with same descriptive statistics as above by cohort and overall.

Mean (±SE) of Ctrough and Ceoi (only for isatuximab) will be plotted over treatment phase by cohort and overall for isatuximab and for atezolizumab.

Individual Ctrough ratio and Ceoi ratio (described in Table 6) will be listed and summarized by descriptive statistics by cohort and overall as described above.

Table 6 - Ctrough and Ceoi ratio

| Analyte | C <sub>trough</sub> | C <sub>eoi</sub> |
|--------------|---------------------|------------------|
| Isatuximab | C2D1 vs C1D1 T168h | C2D1 vs C1D1 |
| | C4D1 vs C1D1 T168h | C4D1 vs C1D1 |
| Atezolizumab | C4D1 vs C2D1 | NA |
| | C8D1 vs C2D1 | NA |

NA = Not applicable.

# 2.4.7.3 Immunogenicity impact on PK

Immunogenicity impact on PK analysis may be explored, depending on the ADA prevalence.

A descriptive statistics of Ctrough as described above will be provided at each cycle in the subset of negative patients by cohort and overall where positive or inconclusive patients will be observed.

A graphical representation of individual Ctrough profile will be provided throughout the course of treatment by cohort and possibly overall where positive or inconclusive patients will be observed. Positive patients profile will be highlighted (eg, color or bold) and the concentration of isatuximab and atezolizumab at the same time as ADA positive result will be notified.

#### 2.4.7.4 Over treatment: population PK approach of isatuximab and atezolizumab

In addition, populations PK approaches may be used for both compounds and PK estimates may be used to conduct exploratory exposure-response analyses for safety and efficacy and PK/PD analyses for relevant biomarkers. If done, the data generated will be reported in stand-alone report(s).

These analyses, if applicable, will be described in the Population Analysis Plan (PAP) which will be issued separately from this Statistical Analysis Plan.

# 2.4.8 Analyses of biomarker variables

The biomarker variables may be summarized by clinical group (eg, SD >6 months vs. others) and overall depending on availability of assessable tumor biopsy samples. Graphics will be provided as appropriate. The biomarker variables include, but not limited to, the following variables:

- CD38 expression.
- PDL1 expression.

Additional biomarker analysis may be conducted in an exploratory manner. Additional analysis, not specified in the protocol but related to the drug action and/or effect of isatuximab/ Atezolizumab, may be conducted on remaining samples pending evolving literature.

# 2.4.9 Analyses of quality of life/health economics variables

Not applicable.

# 2.4.10 Further therapy after discontinuation of investigational medicinal product administration during the study

A listing of further therapy after discontinuation of investigational medicinal product administration during the study may be provided.

#### 2.5 DATA HANDLING CONVENTIONS

# 2.5.1 General conventions

The following formulas will be used for computation of parameters.

# Estimated glomerular filtration (eGRF) using the equation of MDRD formula:

GFR = 
$$175 \times (Scr)^{-1.154} \times (Age)^{-0.203} \times (0.742 \text{ if Female}) \times (1.212 \text{ if African American})$$

with serum creatinine in mg/dL and age in year.

#### Corrected calcium formula:

Corrected Calcium (mmol/L) = Serum Calcium (in mmol/L) + 0.8 (4 - serum albumin [in g/dL])

#### 2.5.2 Data handling conventions for secondary efficacy variables

Not applicable.

#### 2.5.3 Missing data

The analyses and summaries of continuous and categorical variables will be based on observed data only. Percentages will be calculated using as denominator the number of patients with non-missing observation in the considered population. When relevant, the number of patients with missing data is presented.

Property of the Sanofi Group - strictly confidential

When incomplete or missing dates were found in the eCRF, attempts were made to retrieve the complete date, especially for dates within the month prior to first dose. However, if some dates remain incomplete, the following rules will be applied:

# Handling of disease characteristics missing/partial dates

- If the day is missing, it will be estimated by 1.
- If the month is missing, it will be estimated by 1 (only for medical history variables).
- If the year is missing, no estimation will be performed.

# Handling of medication missing/partial dates

No imputation of medication (other than anti-cancer therapies) start/end dates or times will be performed. If a medication date or time is missing or partially missing and it cannot be determined whether it was taken prior or concomitantly, it will be considered a prior, concomitant, and post-treatment medication.

For prior anti-cancer therapies, following rules will be applied:

Missing/partial start date will be imputed as follows:

- If year and month exist, day is missing, impute as the first day of the month.
- If only year exists, month and day are missing, impute as the first day of the year.
- If year, month, and day are all missing, no imputation will be applied.

Missing/partial end date will be imputed in a two-step approach as follows:

- Step 1: Use the following rule to impute end date:
  - If year and month exist, day is missing, impute as the first day of the month,
  - If only year exists, month and day are missing, impute as the first day of the year,
  - If year, month, and day are all missing, no imputation will be applied.
- Step 2: If imputed end date is earlier than start date, set the imputed end date the same as start date.

# Imputation of incomplete date for post anti-cancer treatment start date

For post anti-cancer treatments, if the medication start date is missing, it will be imputed as follows:

- If the medication start day and month are missing and the medication start year is the same as treatment end year, the medication start date will be set equal to treatment end date + 1.
- If the medication start day and month are missing and the medication start year is after the treatment end year, the medication start day and month will each be set to 01.
- If the medication start day is missing and medication start year and month is the same as the treatment end year and month, the medication start day will be set equal to the treatment end day + 1.

Property of the Sanofi Group - strictly confidential

- If the medication start day is missing and medication start month is before the treatment end month and the medication start year is the same as treatment end year, the medication start day will be set to 01.
- If the medication start day is missing and the medication start month is after the treatment end month and the medication start year is the same as treatment end year, the medication start day will be set to 01.
- If the medication start day is missing and the medication start month is not missing and the medication start year is after the treatment end year, the medication start day will be set to 01
- If the medication start day, start month and start year is missing, the medication start date will be set equal to the treatment end date + 1.

No imputation will be done for the missing/partial end date.

# Handling of adverse events with missing or partial date of onset

Missing or partial adverse event onset dates (occurrence or becoming serious) will be imputed so that if the partial adverse event onset date information or visit number does not indicate that the adverse event started prior to treatment or after the treatment-emergent adverse event period, the adverse event will be classified as treatment-emergent. In case of AEs worsening during the study, the emergence will also be based on the cycle of worsening. No imputation of adverse event end dates will be performed. These data imputations are for categorization purpose only and will not be used in listings. No imputation is planned for date of adverse event resolution.

# Handling of death with missing or partial date of death

The imputation for missing or partial death date will proceed as follows:

- If the death day is missing and the death month and year are the same as the last month and year the patient was last known to be alive, the death day will be set equal to the last day the patient was known to be alive + 1.
- If the death day is missing and the death month is after the month the patient was last known to be alive and the death year is the same as the year the patient was last known to be alive, the death day will be set to 01.
- If the death day and month are missing and the death year is the same as the year the patient was last known to be alive, the death date will be set equal to the date the patient was last known to be alive + 1.
- If the death day and month are missing and the death year is after the year the patient was last known to be alive, the death day and month will both be set to 01.

If the date the patient was last known to be alive is partial or missing, no imputation for missing or partial death date will be performed. The last date the patient was known to be alive is the last of: date of last dose, date of last visit performed (when the patient is known to be alive according to subject vital status), date of last laboratory assessment, and date of last vital signs.

# Handling of AEs with missing grade

If the grade is missing for one of the treatment emergent occurrences of an AE, the maximal severity on the remaining occurrences will be considered. If the severity is missing for all the occurrences, no imputation will be done and missing grades will be summarized in the "all grades" category.

# Handling of missing assessment of relationship of adverse events to investigational medicinal product

If the assessment of the relationship to the regimen is missing, then the relationship to the regimen has to be assumed and the adverse event considered as such in the frequency tables of possibly related adverse events, but no imputation should be done at the data level. No imputation will be done for relationship to NMIP.

# Handling of parameters expressed as inequality or approximation

For some parameters (such as laboratory parameters), if the value is expressed as "<xx", "\( \le xx \), half of the numeric portion of the entry or limit of quantification will be used in calculations.

# Handling of missing date/time in duration of infusion calculation

When both atezolizumab and isatuximab are given to a patient on the same visit:

- Missing atezolizumab end date/time will be imputed by isatuximab start date/time (if available).
- Missing isatuximab start date/time will be imputed by atezolizumab end date/time (if available).

Other types of missing date/time will not be imputed, and data will be excluded from the analysis of duration of infusion.

# Handling of other missing dates

Incomplete date of cancer diagnosis:

- If the day of the cancer diagnosis is missing, the date will be imputed to the first day of the month.
- If day and month of the cancer diagnosis are missing, no imputation will be done.

Incomplete date of progression for the last prior regimen:

- If the day of the progression for the last prior regimen is missing, the date will be imputed to the end day of the month.
- If day and month of the progression for the last prior regimen are missing, no imputation will be done.

Incomplete date of prior surgery:

- If the day of the last prior surgery is missing, the date will be imputed to the end day of the month.
- If day and month of the last prior surgery are missing, no imputation will be done.

Incomplete date of prior radiotherapy:

- If the day of the last prior radiotherapy is missing, the date will be imputed to the end day of the month.
- If day and month of the last prior radiotherapy are missing, no imputation will be done.

# 2.5.4 Windows for time points

#### Laboratory data

A protocol planned laboratory test is considered to have occurred during a cycle if the date of sampling is after (>) the first day of the cycle, but prior to or equal ( $\leq$ ) to the first day of the next cycle. For unscheduled tests, a test is considered to have occurred during a cycle if the date of sampling is equal to or after ( $\geq$ ) the first day of the cycle, but prior (<) to the first day of the next cycle.

#### 2.5.5 Unscheduled visits

Unscheduled visit measurements of laboratory data, vital signs and ECG will be used for computation of worst values and/or grades on treatment. Unscheduled visits prior to first administration will be also used for computation of baseline except if they are not collected on the day of first administration.

# 2.5.6 Pooling of centers for statistical analyses

Data from all sites will be pooled together for analyses.

# 2.5.7 Statistical technical issues

Not applicable.

# 3 INTERIM ANALYSIS

An IA for each cohort will be performed for HCC, SCCHN, EOC, and GBM cohorts after the last participants remaining in the treatment period among the first 26, 26, 17 and 31 participants, respectively, in Phase 2 have completed approximately 6 months of study treatment or permanently discontinued both atezolizumab and isatuximab, whichever comes first. The IA may be conducted earlier if the required number of responses for proceeding to Phase 2 Stage 2 is achieved for HCC, SCCHN, and EOC cohorts.

The analysis will include the following parameters/analyses (defined in Section 2.1): RR for patients with HCC or SCCHN or EOC, PFS-6 for patients with GBM, demographics and baseline characteristics, prior or concomitant medication, AEs (TEAE, death, SAE, TEAE leading to discontinuation, IAR, AESI), and laboratory variables (abnormality of hematological and chemistry test). If needed, more data will be analyzed to inform the futility decision including additional efficacy, PK, and biomarker.

# 4 DATABASE LOCK

The database will be locked when clinical review of the database has been completed and all critical queries have been resolved.

# 5 SOFTWARE DOCUMENTATION

All summaries and statistical analyses will be generated using SAS® Version 9.4 or higher.

# 6 REFERENCES

- 1. Eisenhauer EA, Therasse P, Bogaerts J Schwartz LH, Sargent D, Ford R et al. New response evaluation criteria in solid tumours: Revised RECIST guideline (version 1.1). Eur J Cancer. 2009;45:228-47.
- 2. Wen PY, Macdonald DR, Reardon DA, Cloughesy TF, Sorensen AG, Galanis E et al. Updated Response Assessment Criteria for High-Grade Gliomas: Response Assessment in Neuro-Oncology Group. J Clin Oncol. 2010;28(11):1963-72.
- 3. Seymour L, Bogaerts J, Perrone A, Ford R, Schwartz LH, Mandrekar S, et al. iRECIST: guidelines for response criteria for use in trials testing immunotherapeutics. Lancet Oncol. 2017;18:e143-52.
- 4. Okada H, Weller M, Huang R, Finocchiaro G, Gilbert M, Wick W et al. Immunotherapy Response Assessment in Neuro-Oncology (iRANO): a report of the RANO working group. Lancel Oncol. 2015;16(15):e534-42.
- 5. Alexander Kratz, Maryjane Ferraro, Patrick M. Sluss and Kent B. Lewandrowski, MD. Laboratory reference values.

# 7 LIST OF APPENDICES

Appendix A Generic ranges for hematological and biochemistry parameters

# Appendix A Generic ranges for hematological and biochemistry parameters

Table 7 - Generic ranges for hematological parameters

| Test | Gender | Unit | Lower/Upper limit of norma |
|--------------|--------|--------|----------------------------|
| Hemoglobin | F | g/L | 120 - 160 |
| Hemoglobin | М | g/L | 135 - 175 |
| Lymphocytes | | 109/L | 1 - 2 |
| Neutrophils | | 109/L | 1.8 - 3.15 |
| Platelets | | 109/L | 150 - 350 |
| Leukocytes | | 109/L | 4.5 - 11 |
| Eosinophils | | 109/L | 0 - 0.4 |
| Basophils | | 109/L | 0 - 0.15 |
| Monocytes | | 109/L | 0.18 - 0.5 |
| Hematocrit | М | Ratio | 0.41 -0.53 |
| Hematocrit | F | Ratio | 0.36 - 0.46 |
| Erythrocytes | F | 1012/L | 4 - 5.2 |
| Erythrocytes | М | 1012/L | 4.5 -5.9 |
| INR | | ratio | 0.8 -1.2 |

Based on Kratz et al. (5)

Table 8 - Generic ranges for biochemistry parameters

| Test | Unit | Lower – Upper limit of normal |
|--------------------|--------|-------------------------------|
| Albumin | g/L | 35 - 55 |
| BUN | mmol/L | 3.6 - 7.1 |
| Calcium | mmol/L | 2.2 - 2.6 |
| Chloride | mmol/L | 80 - 115 |
| Corrected calcium | mmol/L | 2.2 - 2.6 |
| Glucose | mmol/L | 3.9 - 7 |
| Bicarbonate (HCO3) | mmol/L | 22 - 29 |
| Carbon dioxide | mmol/L | 21 - 30 |
| Potassium | mmol/L | 3.5 - 5 |
| Magnesium | mmol/L | 0.8 - 1.2 |
| Sodium | mmol/L | 136 - 145 |
| Phosphate | mmol/L | 1 - 1.4 |
| Protein | g/L | 55 - 80 |
| Urea | mmol/L | 3.6 - 7.1 |

# Signature Page for VV-CLIN-0549031 v1.0 act15377-16-1-9-sap

| Approve & eSign |
|-----------------|
| Approve & eSign |